CLINICAL TRIAL: NCT05399693
Title: Characterization of Anti-HLA I Antibodies Involved in Platelet Transfusion Refractoriness: Optimization of the Transfusion Management of Patients With Severe Thrombocytopenia
Brief Title: Platelet Transfusion Refractoriness
Acronym: ACERTP
Status: Completed | Type: Observational
Sponsor: Institut de cancérologie Strasbourg Europe (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-006
Record Dates: First submitted 2022-05-25; First posted 2022-06-01 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Platelet Transfusion Refractoriness
MeSH Terms: interventions — Platelet Transfusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Platelet Transfusion Refractoriness
  Interventions: Procedure: platelet transfusion
- Patients without Platelet Transfusion Refractoriness
  Interventions: Procedure: platelet transfusion

INTERVENTIONS:
Procedure: platelet transfusion — platelet transfusion realised for Hematopoietic stem cells graft or for acute leukemia

SUMMARY:
Platelet Transfusion Refractoriness is one of the severe complications after multiple transfusions in patients with severe thrombopenia. Platelet Transfusion Refractoriness is characterized by inefficient transfusion and arise from allo-antibodies specific of platelets antigenes, mostly carried by HLA-I molecules.

DETAILED DESCRIPTION:
A preliminary study has shown different isotypes of anti-HLA I in patients with Platelet Transfusion Refractoriness. Our hypothesis is that the type of anti-HLA I antibodies (recognised epitope, quantity, isotype) should establish predictive and diagnostic criteria for Platelet Transfusion Refractoriness.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient with Hematopoietic stem cells graft (autograft or allograft) or with acute leukemia with the indication of platelet transfusion.

Exclusion Criteria:

* Patient under guardianship
* Minor patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient :
  * with Hematopoietic stem cells graft (autograft or allograft)
  * or with acute leukemia with the indication of platelet transfusion.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2023-08-08 (Actual); Study Completion 2023-08-08 (Actual)

PRIMARY OUTCOMES:
Research of predictive criteria of Platelet transfusion refractoriness | blood samples before the transfusion of each chemotherapy cycle
  Characterisation of anti-HLA I antibodies (recognised epitopes and isotypes) associated to Platelet transfusion refractoriness

CONTACTS AND LOCATIONS:
Overall Officials: Luc FORNECKER, Principal Investigator — Institut de cancérologie Strasbourg Europe
Locations (1):
- Institut de cancérologie Strasbourg Europe, Strasbourg, France

REFERENCES:
- [Derived] Couvidou A, Wald M, Angenieux C, Pires-Marafon J, Apithy MJ, Humbrecht C, Fornecker LM, Congy-Jolivet N, Dupuis A, Rollin J, Maitre B. Anti-HLA class I IgG subclasses skew platelet activation mechanisms in transfusion refractoriness. Haematologica. 2026 Feb 1;111(2):535-545. doi: 10.3324/haematol.2025.287677. Epub 2025 Sep 18. PMID 40963382